CLINICAL TRIAL: NCT02096484
Title: Group Metacognitive Therapy Versus Mindfulness Meditation Therapy in a Transdiagnostic Patient Sample: A Feasibility Study
Brief Title: A Feasibility Study of Group Metacognitive Therapy Versus Mindfulness Meditation Therapy
Acronym: MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical & Experimental Psychopathology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UM145073
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Metacognitive therapy; mindfulness meditation therapy; group therapy; generalized anxiety disorder; Group Based Metacognitive Therapy; Group Based Mindfulness Meditation Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — 2-methylcyclopentadienyl manganese tricarbonyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metacognitive Therapy (Experimental): Individuals randomly assigned to the metacognitive therapy group will undergo group metacognitive therapy for generalized anxiety disorder.. Individuals will undergo 8 sessions of group therapy lasting approximately 90 minutes.
  Interventions: Behavioral: Group Metacognitive Therapy
- Mindfulness Meditation Therapy (Experimental): Individuals randomly assigned to the mindfulness meditation therapy group will undergo group mindfulness meditation therapy for generalized anxiety disorder. Individuals will undergo 8 sessions of group therapy lasting approximately 90 minutes.
  Interventions: Behavioral: Mindfulness Meditation Therapy

INTERVENTIONS:
Behavioral: Group Metacognitive Therapy
  Other Names: MCT
  Arms: Metacognitive Therapy
Behavioral: Mindfulness Meditation Therapy
  Other Names: MMT
  Arms: Mindfulness Meditation Therapy

SUMMARY:
The study will examine the effectiveness of group metacognitive therapy in comparison with group meditation therapy, in patients with Generalised Anxiety Disorder. Individuals will be randomly assigned to either meditation or metacognitive therapy and undergo 8 group therapy sessions of their respective treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* individual's score on the GAD-7 & PHQ-9
* individuals who meet the DSM-IV (Diagnostic and Statistical Manual) criteria for generalized anxiety disorder

Exclusion Criteria:

* Individuals with major depressive disorder
* Individuals who report suicidality
* Individuals with a brain injury or neurological insult
* Individual who currently engage in substance abuse
* Individuals with bipolar disorder
* Individuals with psychotic symptoms
* Individuals who cannot converse or read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Administered at pre treatment, mid treatment, post treatment, and 6 month follow up

SECONDARY OUTCOMES:
CAS-I | Administered at pre treatment, mid treatment, post treatment, and 6 month follow up
GAD-7 | Completed prior to week 1 of treatment.This will be administered prior to treatment as a screening measure for levels of anxiety.
PHQ-9 | Completed prior to week 1 of treatment.This will be administered prior to treatment as a screening measure for levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Capobianco, Principal Investigator — University of Manchester; James Thompson, Principal Investigator — University of Manchester
Locations (1):
- The Rawnsley Building, Manchester Royal Infirmary, Oxford Road, Manchester, Lancashire, United Kingdom